CLINICAL TRIAL: NCT00600977
Title: A Multicentric Phase II-III Randomized Study Safety of Intraveinous Liposomal Pegylated Doxorubicin Versus Continuous Infusion of Doxorubicin During Induction Treatment of Acute Lymphoblastic Leukemia in Patients
Brief Title: Liposomal Anthracyclin in the Treatment of Elderly ALL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: French Innovative Leukemia Organisation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GOELAL LALA SA1; U01-AA1234-01
Record Dates: First submitted 2007-09-26; First posted 2008-01-25 (Estimated); Last update posted 2008-06-26 (Estimated); Status verified 2008-06

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: ALL; Chemotherapy; Pharmacokinetics of doxorubicin (pegylated or not); elderly ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- doxorubicine (Active Comparator): VAD
  Interventions: Drug: Doxorubicine
- Doxorubicine pegylated (Experimental): Doxorubicine pegylated 40 MG/M² J1
  Interventions: Drug: Doxorubicine pegylated

INTERVENTIONS:
Drug: Doxorubicine — 9mg/m² J1 J4 2 COURSES
  Arms: doxorubicine
Drug: Doxorubicine pegylated — 40 MG/M² J1 2 courses
  Arms: Doxorubicine pegylated

SUMMARY:
Phase II multicentric study comparing VAD regimen with continuous infusion over 96 hours of doxorubicin, vincristine and dexamethasone to a 90 minutes infusion of equivalent doses of Dox li-PEG, bolus infusion of vincristine and dexamethasone

DETAILED DESCRIPTION:
Patients aged 55 years or over will be assessed for response to steroids from day -7 to day 0 During steroid therapy, Ph status will be determinated : patients with Ph+ ve ALL will be treated according to the another French Protocol while patients with Ph-ve ALL will be included in the "caelyx" protocol and randomly allocated to induction with VAD or with vadox-li-Peg (caelyx).

A second course of induction therapy with VAD+ cyclophosphamide of Vadox-li-peg+ cyclophosphamide(according to the initial randomization arm) will then be given to all patients.

Consolidation therapy included 2 courses of vad or of vadox-li-Peg , according to the initial random allocation, followed by two courses of cytarabine,cyclophosphamide and thioguanine.

During induction and consolidation therapy, doxorubicin and liposomal pegylated doxorubicin pharmacokinetics will be assessed in all patients.

Treatment of occult CNS invasion includes skull radiotherapy and 6 intrathecal injections(steroÏds+methotrexate) A two years maintenance course with 6 mercaptopurine and methotrexate will then be offered to all patients.

ELIGIBILITY:
Inclusion Criteria:

* 55 years of age and older
* ECOG performance </=2 or >/=3
* VIH negative
* Absence of previous ALL treatment
* Informed consent signed
* SGPT and Bilirubin < 4x upper limit of normal
* Normal creatinine for age
* cardiac state compatible with anthacyclin

Exclusion Criteria:

* ALL with Philadelphia Chromosome
* ALL3
* CML blasts crisis
* Cardiac insufficiency and/ or left ventricular ejection fraction < 50%
* Evolutive infection
* Presence of other evolutifs cancer or ongoing treatment

  * mental status incompatible with inform consent

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2002-03; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Number of patients alive by day 113 ( last injection of anthracycline ) and having received a full course of induction/consolidation therapy | 113 days

SECONDARY OUTCOMES:
Hematological and cutaneous adverse evnts of both types of chemotherapy | 113 days
Resistance to chemotherapy | 113 days
Complete response rates | 113 days
Disease free and overall survival | 4 months
Economical study | 113 days

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde HUNAULT BERGER, RN, Principal Investigator — French Innovative Leukemia Organisation
Locations (1):
- Regional university hospital, Angers, France

REFERENCES:
- [Derived] Hunault-Berger M, Leguay T, Thomas X, Legrand O, Huguet F, Bonmati C, Escoffre-Barbe M, Legros L, Turlure P, Chevallier P, Larosa F, Garban F, Reman O, Rousselot P, Dhedin N, Delannoy A, Lafage-Pochitaloff M, Bene MC, Ifrah N, Dombret H; Group for Research on Adult Acute Lymphoblastic Leukemia (GRAALL). A randomized study of pegylated liposomal doxorubicin versus continuous-infusion doxorubicin in elderly patients with acute lymphoblastic leukemia: the GRAALL-SA1 study. Haematologica. 2011 Feb;96(2):245-52. doi: 10.3324/haematol.2010.027862. Epub 2010 Oct 22. PMID 20971822